CLINICAL TRIAL: NCT00623389
Title: Evaluation of Advanced Lower Extremity Neuroprostheses
Brief Title: Evaluation of an Advanced Lower Extremity Neuroprostheses
Acronym: LE-IST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Ronald J. Triolo, Biomedical Engineer, Case Western Reserve University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EB-001889
Record Dates: First submitted 2008-01-24; First posted 2008-02-26 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Spinal Cord Injuries; Stroke; Paralysis; Tetraplegia; Paraplegia
Keywords: Neurologic disorders; Rare disease; Spinal cord injuries; Stroke; Paraplegia; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Paralysis; Quadriplegia; Paraplegia; Nervous System Diseases; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Implant (Experimental): Volunteers are evaluated for appropriateness for inclusion in the study on an intent-to-treat basis. Qualifying candidates all receive the implanted neuroprosthesis and participate in post-operative training and follow-up procedures.
  Interventions: Device: IST (Implanted Stimulator-Telemeter)

INTERVENTIONS:
Device: IST (Implanted Stimulator-Telemeter) — Pre-surgical exercise with surface electrical stimulation, surgery including electrode and IST- implanted pulse generator insertion, exercise and physical therapy with the implanted system, functional training and laboratory assessment of clinical and technical performance.

SUMMARY:
The purpose of this study is to evaluate a surgically implanted functional electrical stimulation (FES) system to facilitate exercise, standing, stepping and/or balance in people with various degrees of paralysis.

DETAILED DESCRIPTION:
Protocol Outline: Patents undergo surgery in which electrodes are implanted into muscles of the trunk and legs. Electrode leads are connected to an stimulator/telemeter. Following implantation, patients undergo training in standing, transfers and other advanced mobility skills using the functional electrical stimulation system. A prescribed course of exercise, functional training and rehabilitation with the implanted stimulation system, followed by laboratory assessments of strength, balance and functional abilities with and without the system, as well as the technical performance of the implanted components. Home-based training follows prior to discharge for home use of the system.

Patients are followed at 6 and 12 months after discharge and then annually thereafter.

ELIGIBILITY:
Phase I Inclusion Criteria

1. Skeletal maturity and ability to sign informed consent (>18 years)
2. Non-ventilator dependent paralysis resulting from injuries such as: mid cervical/thoracic (C4 or below) spinal cord injuries, poststroke hemiparesis, TBI, or MS, affecting the trunk and/or lower limbs
3. Innervated and excitable lower extremity and trunk musculature
4. Adequate social support and stability
5. Willingness to comply with follow-up procedures

Phase I Exclusion Criteria

1. Non-English speaking
2. Females who are pregnant
3. Current pressure injuries that would be exacerbated by study activities
4. Severe contractures or uncontrolled spasticity of any major joint of the upper or lower extremities that results in a fixed deformity that would interfere with study activities
5. History of spontaneous fractures or other evidence of excessively low bone density
6. History of vestibular dysfunction, balance problems, or spontaneous falls
7. Acute and or/untreated orthopedic problems that would prevent a participant from weight bearing or exercising such as a dislocation or fracture.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Device reliability and technical performance measuring changes in standing duration from baseline at discharge to 12 months after discharge | Change from immediately after intervention and 1 year after intervention
  Repeated measures of standing duration in minutes
Device reliability and technical performance measuring changes in standing loads from baseline at discharge to 12 months after discharge | Change from immediately after intervention and 1 year after intervention
  Repeated measures of arm/leg loading measured in Kg
Device reliability and technical performance measuring changes in walking distance from baseline at discharge to 12 months after discharge | Change from immediately after intervention and 1 year after intervention
  Repeated measures of walking distance in meters
Device reliability and technical performance measuring changes in walking duration from baseline at discharge to 12 months after discharge | Change from immediately after intervention and 1 year after intervention
  Repeated measures of walking time in minutes

SECONDARY OUTCOMES:
Device operability measuring changes in functional activities of daily living from baseline at discharge and 12 months after discharge | Change from immediately after intervention and 1 year after intervention
  Repeated measures of standing reach in cm, and transfer height in cm

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Triolo, Ph.D., Principal Investigator — Case Western Reserve University; Musa L Audu, Ph.D., Principal Investigator — Louis Stokes Cleveland VA Medical Center
Locations (2):
- United States (2):
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - MetroHealth System, Cleveland, Ohio

REFERENCES:
- [Background] Fisher LE, Miller ME, Nogan SJ, Davis JA, Anderson JS, Murray LM, Tyler DJ, Triolo RJ. Preliminary evaluation of a neural prosthesis for standing after spinal cord injury with four contact nerve-cuff electrodes for quadriceps stimulation. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:3592-5. doi: 10.1109/IEMBS.2006.260833. PMID 17947042
- [Background] Dutta A, Kobetic R, Triolo RJ. Ambulation after incomplete spinal cord injury with electromyogram-triggered functional electrical stimulation. Conf Proc IEEE Eng Med Biol Soc. 2006;2006:5408-11. doi: 10.1109/IEMBS.2006.259257. PMID 17946304
- [Background] Mushahwar VK, Jacobs PL, Normann RA, Triolo RJ, Kleitman N. New functional electrical stimulation approaches to standing and walking. J Neural Eng. 2007 Sep;4(3):S181-97. doi: 10.1088/1741-2560/4/3/S05. Epub 2007 Aug 22. PMID 17873417
- [Background] Uhlir JP, Triolo RJ, Davis JA Jr, Bieri C. Performance of epimysial stimulating electrodes in the lower extremities of individuals with spinal cord injury. IEEE Trans Neural Syst Rehabil Eng. 2004 Jun;12(2):279-87. doi: 10.1109/TNSRE.2004.827224. PMID 15218941
- [Background] Bogie KM, Triolo RJ. Effects of regular use of neuromuscular electrical stimulation on tissue health. J Rehabil Res Dev. 2003 Nov-Dec;40(6):469-75. doi: 10.1682/jrrd.2003.11.0469. PMID 15077659
- [Background] Agarwal S, Triolo RJ, Kobetic R, Miller M, Bieri C, Kukke S, Rohde L, Davis JA Jr. Long-term user perceptions of an implanted neuroprosthesis for exercise, standing, and transfers after spinal cord injury. J Rehabil Res Dev. 2003 May-Jun;40(3):241-52. PMID 14582528
- [Background] Davis JA Jr, Triolo RJ, Uhlir J, Bieri C, Rohde L, Lissy D, Kukke S. Preliminary performance of a surgically implanted neuroprosthesis for standing and transfers--where do we stand? J Rehabil Res Dev. 2001 Nov-Dec;38(6):609-17. PMID 11767968
- [Derived] Triolo RJ, Bailey SN, Foglyano KM, Kobetic R, Lombardo LM, Miller ME, Pinault G. Long-Term Performance and User Satisfaction With Implanted Neuroprostheses for Upright Mobility After Paraplegia: 2- to 14-Year Follow-Up. Arch Phys Med Rehabil. 2018 Feb;99(2):289-298. doi: 10.1016/j.apmr.2017.08.470. Epub 2017 Sep 9. PMID 28899825